CLINICAL TRIAL: NCT06606080
Title: The Formation Pathway of Fear of Cancer Recurrence in Gastric Cancer Survivors From a Time Perspective
Brief Title: The Relationship Between Time Perspective, Fear of Cancer Recurrence, Rumination, and Catastrophizing in Gastric Cancer Survivors
Status: Completed | Type: Observational
Sponsor: Ting Wang (Other)
Responsible Party: Sponsor-Investigator, Ting Wang, Principal Investigator, Nanjing Medical University
Organization: Nanjing Medical University (Other)
Other Study IDs: 2023540
Record Dates: First submitted 2024-09-17; First posted 2024-09-20 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Gastric Cancer Patient

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The temporal perspective provides a theory oriented to temporal insights that can shed light on the role of cognitive coping styles in the formation of fear of cancer recurrence. The self-regulatory executive function model elucidates the central role of rumination thinking, catastrophizing cognitive coping styles in the formation of cancer recurrence fear. Therefore, this study will rely on both theoretical models to construct a cognitive appraisal coping model to explore the formation pathway of cancer recurrence fear

ELIGIBILITY:
Inclusion Criteria:

* Preoperative gastroscopy and pathological diagnosis of gastric cancer;
* Aged 18 years or older
* There is no history of recurrent disease or new primary cancer
* Received surgical resection of cancerous tissues or radiotherapy treatment
* Conscious, with normal communication and comprehension ability
* The patients were aware of their own condition and diagnosis, and informedly agreed to participate in this study

Exclusion Criteria:

● History of mental or cognitive impairment prior to cancer diagnosis

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Select elderly gastric cancer patients who were receiving medical treatment at a tertiary hospital
Sampling Method: Probability Sample
Enrollment: 340 (Actual)
Dates: Start 2023-08-10 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-10 (Actual)

PRIMARY OUTCOMES:
Time perspective | through study completion, an average of 1 year
  The Chinese version of ZIPI scale was adopted for the measurement of time perspective, ZIPI scale is the current international common measurement tool.ZTPI scale was developed by Zimbardo et al. in 1999, which is mainly used for assessing individual's time perspective, the scale has been translated by scholars from many countries, and has good cross-cultural applicability. The Chinese version of the ZTPI scale was Chineseized and revised by Wang Chen in 2016, and the revised scale can be divided into five dimensions of past negativity (7 entries), past positivity (6 entries), present impulsivity (4 entries), future (5 entries), and present predestination (3 entries), with a total of 25 entries after exploratory factor analysis.All questions are scored on a scale of 1 (strongly disagree) to 5 (strongly agree), with higher scores indicating a greater tendency towards certain time perspective.
Catastrophizing | through study completion, an average of 1 year
  Catastrophizing was measured using the 4-item Cognitive Emotion Regulation Questionnaire Catastrophizing subscale ( CERQ-CS ). Chinese scholars such as Zhu Xiongzhao (2007) revised the Cognitive Emotion Regulation Questionnaire (CERQ) to form the Chinese version of the Cognitive Emotion Regulation Questionnaire (CERQ-C) applicable to the Chinese version.Each item of the CERQ - CS has 5 responses ranging from 1 (almost never) to 5 (almost always). Higher total scores on this subscale indicate higher levels of catastrophizing, and this subscale has good reliability in the Chinese population, the minimum value is 4 points, and the maximum value is 20 points
Rumination | through study completion, an average of 1 year
  Intrusive rumination was measured using the Event-Related Rumination Rumination Questionnaire (ERRI). It is scored according to how many rumination the subjects have produced in the last two weeks and the number of scores is used to assess the degree of rumination of the individual. It was revised by Zhou Xiao et al. (2014) to Cann et al.'s (2010) Event-Related Rumination Questionnaire, which included two dimensions of intrusive rumination and active rumination, with a total of 20 questions. After the revision, the questionnaire had good internal consistency coefficients for the total and dimensions, and the validity indicators also reached a good level. Each item is rated on a 4 point scale, and the scores of the Intrusive rumination scales range from 0 to 30 points The higher the score, the higher the level of invasive rumination.
Fear of cancer recurrence | through study completion, an average of 1 year
  The Chinese version of the Fear of Disease Progression Simplified Scale (FoP-Q-SF) was used to measure the degree of fear of recurrence in cancer patients. Our researchers and scholars, Wu Qiyun et al. translated and Chineseized the FoP-Q-SF according to Chinese characteristics to form a version of the Fear of Progression of Disease Simplified Scale suitable for cancer patients in China. There are 12 questions in total, the higher the score, the higher the level of fear of recurrence. When the score is between 12 and 23, it indicates that the patient is at a low level of fear recurrence. When the score is between 24 and 36, it indicates that the patient is at a moderate level of fear recurrence. When the score is between 36 and 60, it indicates that the patient is at a high level of fear recurrence.

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No